CLINICAL TRIAL: NCT02181452
Title: Evaluation of SWE Performances for the Non-Invasive Diagnosis of Liver Fibrosis in Patients With Chronic Liver Diseases
Brief Title: Liver Fibrosis Assessment With ShearWave Elastography
Status: Completed | Type: Observational
Sponsor: SuperSonic Imagine (Industry)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LE1
Record Dates: First submitted 2014-06-19; First posted 2014-07-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Liver Fibrosis
Keywords: liver; fibrosis; ShearWave Elastography; ultrasound
MeSH Terms: conditions — Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic liver disease/fibrosis can be the result of various causes, and the result is that the liver tissue becomes stiff. ShearWave™ elastography, available on the Aixplorer® ultrasound system, is a method that can be used to measure the stiffness of organs in the body, for example the liver.

This study will evaluate how this technology performs as a non-invasive test to stage liver fibrosis in patients with chronic liver disease.

DETAILED DESCRIPTION:
The measurements of liver stiffness made by the Aixplorer® will be compared to (where available) :

* blood markers
* biopsy results
* other stiffness measurement exams (FibroScan, ARFI, ElastPQ...)

The influence of other (confounding) factors on the reliability of SWE measurements will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting a single condition below:

  * Chronic hepatitis B, defined by serology HBsAg positive and the presence of DNA / RNA in the serum, or
  * Chronic hepatitis C, defined by serology anti-HCV positive and the presence of DNA / RNA in the serum, or
  * non-alcoholic fatty-liver disease
* And meeting all of the conditions below:

  * liver biopsy for histological evaluation of liver fibrosis
  * Length of liver biopsy ≥ 15 mm paraffin sections (except if cirrhosis)
  * Age of majority in their country
  * Obtaining the signature of consent for participation in the data collection, in addition to the routine consent form routinely used at the sites.

Exclusion Criteria:

* Cause of chronic liver disease other than viral (alcohol, hemochromatosis, autoimmune hepatitis, biliary tract disease intrahepatic...) and other than non-alcoholic fatty-liver disease
* History of antiviral therapy for 6 months or less of current antiviral therapy
* Any systemic, viral hepatitis and HIV co-infection
* Pregnant woman
* Failure to obtain consent
* Length of all liver biopsy specimens below 15mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population will consist of patients who have confirmed or suspected liver fibrosis and will be assessed with ultrasound, +/- blood analysis, +/- other non-invasive imaging, and/or measurements, and biopsy
Sampling Method: Non-Probability Sample
Enrollment: 2333 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Correlation coefficients between factors and liver stiffness | Within one year of the study start date
  Factors include patient's clinical and biological parameters

SECONDARY OUTCOMES:
Technical success rates depending on factors | Within one year of the study start date
  Factors include patient's clinical and biological parameters
Diagnostic performance of multivariate models to assess liver fibrosis levels | Within one year of the study start date
  Determined by histological examination of liver biopsy. The resulting tests will be compared on the basis of their AUROC and test of statistical differences.
  Fibrosis levels involved are:
  * at least significant fibrosis (Metavir score F≥2)
  * at least severe fibrosis (Metavir score F≥3)
  * liver cirrhosis (Metavir score F=4)
Sensitivity, specificity, positive and negative predictive values of the best multivariate model to assess liver fibrosis | Within one year of the study start date
  This will be determined by histological examination of liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Freidrich-Rust, Principal Investigator — Johan Goethe University
Locations (13):
- University of Antwerp, Edegem, Belgium
- 3rd Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China
- Odense University Hospital, Odense, Denmark
- France (4):
  - University Hospital of Bordeaux, Bordeaux
  - Beaujon Hospital, Clichy
  - Hopital Edouard Herriot, Lyon
  - Cochin Hospital, Paris
- Germany (2):
  - University of Bonn, Bonn
  - Johan Goethe Universitat, Frankfurt
- University of Athens Medical School, Athens, Greece
- Chinese University of Hong Kong - Prince of Wales Hospital, Hong Kong, Hong Kong
- University of Pavia, Pavia, Italy
- University of Timosoara, Timișoara, Romania